CLINICAL TRIAL: NCT05489133
Title: Early Intervention After Rape to Prevent Post-traumatic Stress Disorder - a Multicenter Randomized Control Trial
Brief Title: Early Psychological Intervention After Rape
Acronym: EIR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other); The Research Council of Norway (Other); Norwegian Women's Public Health Association (Norske Kvinners Sanitetsforening) (Unknown); National Centre for Emergency Primary Health Care, NORCE (Unknown); UiT The Arctic University of Norway (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 348496
Record Dates: First submitted 2022-07-15; First posted 2022-08-05 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Post Traumatic Stress Disorder; Rape Sexual Assault; Sexual Dysfunctions, Psychological; Pelvic Floor Myalgia; Pelvic Pain Syndrome; Depression, Anxiety; Sleep Disturbance; Activity, Motor; Cortisol Deficiency
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Sexual Dysfunctions, Psychological; Vaginismus; Depression; Anxiety Disorders; Parasomnias; Motor Activity | interventions — Crisis Intervention; Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Primary objective is to test whether a psychological intervention with modified prolonged exposure (mPE) therapy is superior to treatment as usual (TAU) to prevent the development of PTSD.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified prolonged exposure (add on) (Experimental): The psychological intervention modified Prolonged Exposure Therapy (mPE) is applied, in addition to Treatment as usual (TAU) (that is, an Add-on). mPE is a trauma-focused evidence-based cognitive behavioral therapy (CBT) shown to be effective in treating PTSD. We will use imaginal exposure in the sessions with the patient describing the traumatic event in detail while being recorded for later listening and homework, and in vivo exposure for visiting specific places or people. Psychoeducation and controlled breathing exercises play a secondary role in PE. We have adapted the mPE to the current SAC settings in Norway where nurses or social workers, not psychologist, as a rule are performing the psychosocial follow-up for rape victims. In this project we plan for three to five once or twice weekly nurse-/social worker-led mPE interventions, given early after the assault.
  Interventions: Behavioral: Modified prolonged exposure
- Treatment as usual (TAU) (No Intervention): Standard care at the sexual assault center (SAC), that is mostly nurse-/social worker-led psychoeducation at varying intervals and extent, and medical follow-up at the SAC.

INTERVENTIONS:
Behavioral: Modified prolonged exposure — Imaginary and in vivo expo, in addition to psychoeducation
  Other Names: Brief intervention; cognitive behavioral therapy
  Arms: Modified prolonged exposure (add on)

SUMMARY:
Rape is a common cause of post-traumatic stress disorder (PTSD) among women, as around 30-50% will develop PTSD in the aftermath of rape. A modified protocol based on Prolonged Exposure Therapy (mPE), has been developed, consisting of three to five once or twice weekly 60 minutes sessions, and studies indicate that if implemented early after rape, mPE may prevent the development of PTSD. The aim of the study is to conduct a multi-site (4 Sexual assault care centers in Norway) randomized control trial (RCT) in which patients are recruited early after rape, and randomized to intervention (mPE) or treatment as usual (TAU).

DETAILED DESCRIPTION:
Rape is a common cause of post-traumatic stress disorder (PTSD) among women, as around 30-50% will develop PTSD in the aftermath of rape, leading to severe mental and physical suffering. There is a lack of evidence-based knowledge how to prevent the development of PTSD after rape. Women may suffer from PTSD for years before receiving therapy.

Prolonged Exposure Therapy (PE) is well documented as a therapy. However, preventing the development of PTSD have the potential to spare women of the suffering, prevent both mental and somatic health problems, and also reduce health care costs. Currently a brief protocol based on PE, has been developed, modified prolonged exposure (mPE), consisting of three to five once or twice weekly 60 minutes sessions, and studies indicate that if implemented early after rape, mPE may prevent the development of PTSD.

Specialized services for victims, Sexual Assault Care (SAC) centers have been established in Norway, offering forensic documentation, medical treatment and psychosocial follow-up. The follow-up service varies widely and no evidence-based preventive measures have been implemented.

The investigators propose to conduct a multi-site (SAC centers in Trondheim, Oslo, and Sandefjord) randomized control trial (RCT) in which patients are recruited early after a rape, and randomized within 2 weeks to intervention (mPE) or treatment as usual (TAU).

The patients will be stratified by treatment center and randomized in permuted blocks of varying sizes according to a computer-generated randomization key prepared by the Clinical Research Unit at .

Around 800 patients will attend one of the four SACs per year. Based on experience from others the investigators anticipate that approximately 200 patients will be eligible and consenting to participation in this study and that around 50% of participants will dropout during the study period. A final sample size of 100 completed participants (50 in the intervention and 50 in TAU) will achieve 80% power to detect a standardized mean difference (SMD) of 0.44 for each of the primary outcomes in a design with 3 repeated measurements assuming an autoregressive, AR(1), covariance structure when the standard deviation is 1, the correlation between observations on the same subject is 0.5, and the alpha level is 0.05 (PASS Sample Size software - Tests for Two Means in Repeated Measures Design). Given the rather conservative estimate for inclusion, the investigators will need 1.5-2 years to recruit sufficient numbers.

Given the nested structure of the data - e.g., multiple measurement points nested within patients, patients nested within therapists, therapists nested within study sites - data will be analyzed by multilevel modeling. In addition, multilevel modeling is a robust method to deal with the missing data given the expected high percentage of drop-out from the study. The primary analysis will be an intention-to-treat analysis.

Predictors and moderators of the intervention, like stress response (measured by level of cortisol in hair and saliva) and sleep patterns (measured with actigraphy), will be explored.

The planned intervention is a brief and simple program, with large potential to be implemented as routines if proven effective, and thus inform clinical guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥ 16 years of age
* attending after a trauma meeting the DSM V trauma definition criterion "sexual violation" (in this context, characterized by penetration in any body orifice, by penis, finger, foreign body, but also attempted penetration leading to a sufficient mental reaction, helplessness, without control, intense fear etc.)

Exclusion Criteria:

* Age < 16 years
* male biological gender
* cognitive disability
* acute psychosis
* acute suicidal
* severe alcohol/drug abuse
* current treatment for PTSD
* non-Norwegian speaking
* total amnesia for the event

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Many of the vaildated questionnaires are based on the presence of female genital organs, hence, we have chosen to include only genetical and phenotypical females
Enrollment: 200 (Estimated)
Dates: Start 2022-06-14 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
PTSD Checklist for DSM-5 (PCL-5) | At 3 months follow-up
  The PCL-5 is a self-report questionnaire consisting of 20 items corresponding to the 20 symptoms of PTSD as defined by DSM-5. Patients rate their posttraumatic symptoms on a Likert scale from 0-4. The continuous sum score of the PCL-5 will de the primary outcome.
PTSD Symptom Scale - Interview for DSM-5 (PSS-I-5) | At 3 months follow-up
  The PSS-I-5 is a clinician-administered diagnostic interview measuring the 20 symptoms of PTSD as defined by DSM-5.

SECONDARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | At 6 weeks, 3, 6 and 12 months
  The PHQ-9 is a self-report questionnaire consisting of nine items measuring the severity of depressive symptoms.
General Anxiety Disorder-7 (GAD-7) | At 6 weeks, 3, 6 and 12 months
  GAD-7 is a self-report questionnaire consisting of seven items measuring the severity of symptoms of anxiety.
Female Sexual Function Index (FSFI) | At 6 weeks, 3, 6 and 12 months
  The FSFI is a multidimensional self-report instrument for the assessment of female sexual function. It contains 19 items divided into six subscales, and gives a total score of 2-36 by multiplying the sum of each subscale with a factor. Mapi Research Trust, a non-profit, full-service provider, promoting the use of Clinical Outcomes Assessments (COAs) have given us permission to use the Norwegian version of the FSFI questionnaire in our study, a version we consider better than the one available on the FHI web-pages.
Bergen insomnia scale (BIS) | At 6 weeks, 3, 6 and 12 months
  Insomnia, questionnaire, quantitative, continous measure. The questionnaire contains 6 items relating to sleep and tiredness. Score 0 -7 (0 means no days during the course of a week, 7 means every day during the course of a week) on each item are summarized.
  Diagnostics for Insomnia: score ≥ 3 on at least one of the items 1 -4, and score ≥ 3 on at least one of the items 5-6) vs. No insomnia: score ≤ 2 on all items 1-4 or score ≤ 2 on both items 5-6
EQ-5D-5L | At 6 weeks, 3, 6 and 12 months
  Quality of life: five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems (each scored 1-5).
  Included also is the EQ VAS that records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine' (0-100). The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement.
The Amsterdam Hyperactive Pelvic Floor Scale for Women | At 6 weeks, 3, 6 and 12 months
  Questionnaire, translated and validated Norwegian version: The original questionnaire includes 30 items. Each item deals with one symptom and has a 5-point Likert scale varying from never (score 1) to very often (score 5). 25 of the 30 items are categorized into six different subscales: 1) vulvar pain symptoms; 2) abdominal pain and defecation symptoms; 3) micturition problems; 4) urinary tract infection; 5) rectal problems; and 6) physiological symptoms of general stress/tension.
  A total score is given from 6 to 30 where a low score (6,0 - 10,9) means "no hyperactivity" in the pelvic floor muscles, a medium score (11,0 - 12,9) means "mild hyperactivity" in the pelvic floor and a high score (13,0 - 30,0) means "moderate to severe hyperactivity" in the pelvic floor.
PTSD Checklist for DSM-5 (PCL-5) | At 6 weeks, 3, 6 and 12 months
  The PCL-5 is a self-report questionnaire consisting of 20 items corresponding to the 20 symptoms of PTSD as defined by DSM-5. Patients rate their posttraumatic symptoms on a Likert scale from 0-4. The continuous sum score of the PCL-5 will de the primary outcome.
PTSD Symptom Scale - Interview for DSM-5 (PSS-I-5) | At 6 weeks, 3, 6 and 12 months
  The PSS-I-5 is a clinician-administered diagnostic interview measuring the 20 symptoms of PTSD as defined by DSM-5.

CONTACTS AND LOCATIONS:
Overall Officials: Cecilie T Hagemann, Principal Investigator — St. Olavs Hospital; Joar Ø Halvorsen, Study Director — St. Olavs Hospital
Locations (4):
- Norway (4):
  - Overgrepsmottaket Sør-Rogaland, Stavanger, In
  - Oslo Emergency Medical Agency (Oslo kommune, Legevakten, Overgrepsmottaket i Oslo), Oslo
  - Sandefjord Emergency Medical Agency (Legevakten, Overgrepsmottaket i Vestfold), Sandefjord
  - Department of Obstetrics and Gynecology, St. Olavs hospital (Overgrepsmottaket), Trondheim

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Haugen T, Halvorsen JO, Friborg O, Mork PJ, Mikkelsen G, Schei B, Hagemann C. Early Intervention after Rape to prevent post-traumatic stress symptoms (the EIR-study): an internal pilot study of a randomized controlled trial. Pilot Feasibility Stud. 2024 Sep 2;10(1):118. doi: 10.1186/s40814-024-01541-0. PMID 39223617
- [Result] Haugen T, Halvorsen JO, Friborg O, Simpson MR, Mork PJ, Mikkelsen G, Elklit A, Rothbaum BO, Schei B, Hagemann C. Modified prolonged exposure therapy as Early Intervention after Rape (The EIR-study): study protocol for a multicenter randomized add-on superiority trial. Trials. 2023 Feb 21;24(1):126. doi: 10.1186/s13063-023-07147-w. PMID 36810120
- [Derived] Haugen T, Halvorsen JO, Friborg O, Schei B, Hagemann CT, Kjelsvik M. Therapists perspectives on the Early Intervention after Rape study: a qualitative process evaluation of a randomized controlled trial. Eur J Psychotraumatol. 2025 Dec;16(1):2443279. doi: 10.1080/20008066.2024.2443279. Epub 2025 Jan 7. PMID 39773406